CLINICAL TRIAL: NCT00091533
Title: Neural Correlates of Observation of Tactile Stimulation in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040278; 04-N-0278
Record Dates: First submitted 2004-09-09; First posted 2004-09-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-09-02

CONDITIONS: Healthy
Keywords: fMRI; Mirror Neuron System; Bimodal Neurons; Somatosensory Cortex; Rehabilitation; Healthy Volunteer; HV

SUMMARY:
This study will examine activity in the brain during the observation of touch. Studies with animals have shown that mirror neurons, or nerve cells, are active during the observation and performance of an action. The researchers for this study hypothesize that a similar system pertains to observing and experiencing touch.

Patients ages 18 to 75 years old who are in good health, are right handed, and who are able to perform simple tasks that require attention may be eligible for this study. Pregnant women are not eligible.

Patients who have not had a health screening at NIH will undergo a clinical and neurological exam. Women of childbearing potential will also have a pregnancy test. The screening will take about 2 to 3 hours. A diagnostic magnetic resonance imaging (MRI) scan will be performed if patients have not undergone one in the previous 12 months. During the procedure, patients will lie still on a table that will slide into the enclosed tunnel of the scanner. They will be asked to lie as still as possible for up to a few minutes at a time. As the scanner takes pictures, patients will hear knocking or beeping sounds, and they will wear earplugs to reduce the noise. Patients will be able to communicate with the MRI staff at all times during the scan, and they may ask to be moved out of the machine at any time. This scan will take about 2 hours.

Two sessions are involved in the study. The first one is intended to familiarize patients with the procedure. During it, they will learn about hand stimulus, through watching a video showing the index finger of a hand being touched by a stick repeatedly. Then the activity will be repeated, but this time, a researcher will also touch the patient's index finger while he or she is watching the video. This session will take about 1 hour.

The second session consists of a functional MRI scan, or fMRI. During it, pictures of the brain will be taken while patients perform tasks. All tasks will be explained in advance, and patients will have an opportunity to practice them before entering the scanner. The fMRI scan will take 1 to 2 hours.

The researchers will discuss the results of the tests with the participants. There is not a direct benefit to those who take part in the study. However, it is hoped that resulting information will enhance researchers' understanding about how the brain processes observed information.

DETAILED DESCRIPTION:
Objective:

There is growing evidence that a mirror system for action observation exists. Neurons in the monkey premotor cortex discharge with performance of goal directed actions and also with observation of another individual performing a similar action. This mirror neuron system for action observation seems to be important for the recognition and understanding of actions. Recently, bimodal neurons, sensitive both for tactile stimulation and for visual stimuli, were found in the parietal cortex. This suggests the idea that there might be a similar mirror neuron system for observing and receiving (or experiencing) tactile stimulation. The neuronal correlates of observing tactile stimulation are mainly unknown. The purpose of this protocol is to determine the pattern of brain activation related to the observation of a tactile stimulated hand.

Study Population:

We will test our hypothesis by means of a functional MRI (fMRI) experiment in a group of healthy subjects.

Design:

We hypothesize that observation of touch will rely on the activation of a cortical network that is different form the observation of non-touch and is in part overlapping with cortical structures active during real tactile stimulation (i.e., somatosensory cortex). Further, we hypothesize that the observation of touch enhances activation in the somatosensory cortex during real tactile stimulation.

Outcome Measures:

Our outcome measure will be an increase in the number of activated voxels in the somatosensory cortex during the touch observation (for both hypothesis). This would give an important hint for a mirror system for observed and received touch. A mirror neuron system for observed touch may become an important tool in rehabilitative treatment for patients with somatosensory impairments.

ELIGIBILITY:
* INCLUSION CRITERIA:

Only healthy right-handed volunteers aged 18 to 75 years who fulfill the inclusion criteria will be included in this protocol.

Subjects should be able to sustain attention to the task over 10 minutes.

All volunteers should have no history of neurological and psychiatric illness.

EXCLUSION CRITERIA:

Volunteers with history of severe alcohol or drug abuse, psychiatric illness like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 23 or less).

Volunteers with severe uncontrolled medical problems (e.g. cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others).

Volunteers with increased intracranial pressure (as evaluated by clinical examination).

Volunteers with unstable cardiac arrhythmia.

Volunteers with history of hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system.

Volunteers with more than moderate to severe microangiopathy (as assessed by multiple peri-ventricular T2 hyperintensity on the pre-experimental anatomical MRI), polyneuropathy (as assessed by clinical examination), diabetes mellitus (medical record), or ischemic peripheral disease (as assessed by clinical examination).

Volunteers who are on medication with the potential to influence nervous system function, who have a history of surgery with metallic implants or a known history of metallic particles in the eye, a cardiac pacemaker, intracardiac lines, neural stimulators, cochlear implants.

Volunteers who are pregnant.

Volunteers with significant visual loss/deficits.

Volunteers with MRI contraindications.

Volunteers with impaired sensation or neuropathy of the hand.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-09-03; Study Completion 2008-09-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Avikainen S, Forss N, Hari R. Modulated activation of the human SI and SII cortices during observation of hand actions. Neuroimage. 2002 Mar;15(3):640-6. doi: 10.1006/nimg.2001.1029. PMID 11848707
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303
- [Background] Fadiga L, Fogassi L, Pavesi G, Rizzolatti G. Motor facilitation during action observation: a magnetic stimulation study. J Neurophysiol. 1995 Jun;73(6):2608-11. doi: 10.1152/jn.1995.73.6.2608. PMID 7666169